CLINICAL TRIAL: NCT04481087
Title: Clinical Comparison of Different Adhesives in NCCLs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCCLs universal
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Tooth Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Clearfil Universal Bond Quick, self-etch mode (CU-SE) (Experimental)
  Interventions: Device: Clearfil Universal Bond Quick
- Clearfil Universal Bond Quick, selective etch mode (CU-SLE) (Experimental)
  Interventions: Device: Clearfil Universal Bond Quick
- Clearfil Universal Bond Quick, etch&rinse mode (CU-ER) (Experimental)
  Interventions: Device: Clearfil Universal Bond Quick
- Clearfil SE Bond (CSE) (Experimental)
  Interventions: Device: Clearfil SE Bond
- Tetric N-Bond (TB) (Experimental)
  Interventions: Device: Tetric N-Bond

INTERVENTIONS:
Device: Clearfil Universal Bond Quick — Adhesive systems
  Arms: Clearfil Universal Bond Quick, self-etch mode (CU-SE)
Device: Clearfil Universal Bond Quick — Adhesive systems
  Arms: Clearfil Universal Bond Quick, selective etch mode (CU-SLE)
Device: Clearfil Universal Bond Quick — Adhesive systems
  Arms: Clearfil Universal Bond Quick, etch&rinse mode (CU-ER)
Device: Clearfil SE Bond — Adhesive systems
  Arms: Clearfil SE Bond (CSE)
Device: Tetric N-Bond — Adhesive systems
  Arms: Tetric N-Bond (TB)

SUMMARY:
The aim of this randomized, controlled, prospective clinical trial is to evaluate the performances of a universal adhesive in three different application modes, a self-etch adhesive and an etch&rinse adhesive in restoration of non-caries cervical lesions. Thirty-four patients will receive restorations. Lesions will be divided into 5 groups according to adhesive systems and application modes: CU-SE: Clearfil Universal Bond Quick in self-etch mode, CU-SLE: Clearfil Universal Bond Quick in selective etch mode, CU-ER: Clearfil Universal Bond Quick in etch&rinse mode, CSE: Clearfil SE Bond, TB: Tetric N-Bond. Restorations (Tetric N-Ceram composite) will be scored with regard to retention, marginal discoloration, marginal adaptation, recurrent caries and post operative sensitivity using modified USPHS criteria after 48 months. Two examiners who is not involved in the placement of restorations will conduct the evaluations. Descriptive statistics will be performed using Chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older,
* having no medical or behavioral problems preventing then from attending review visits,
* having at least 5 tooth with NCCLs
* having antagonist teeth

Exclusion Criteria:

* poor gingival health,
* uncontrolled, rampant caries,
* bruxism,
* removable partial dentures,
* xerostomia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Clinical performances of different adhesives | two years
  Two year examinations according to USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)